CLINICAL TRIAL: NCT02229331
Title: Biomechanical Determinants and Patterns Associated to the Pathophysiological Cascade of Ankle Arthropathy in Children With Haemophilia: Non-invasive In-vivo Measurement of Foot Joints in Children With Haemophilia During Gait.
Acronym: 3DMKFM
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Kevin Deschamps, Dr, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: 3DMKFM_haemo1
Record Dates: First submitted 2014-08-26; First posted 2014-09-01 (Estimated); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Haemophilia; Arthropathy
Keywords: haemophilia; arthropathy; pediatrics; ankle; biomechanics
MeSH Terms: conditions — Hemophilia A; Joint Diseases | interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- gait analysis: gait analysis
  Interventions: Other: Gait analysis

INTERVENTIONS:
Other: Gait analysis

SUMMARY:
Haemophilia is a rare X chromosome-linked coagulation disorder resulting from a congenital deficiency or absence of circulating factor VIII (Haemophilia A) or factor IX (Haemophilia B).As a consequence, patients with haemophilia are unable to generate adequate thrombin resulting in abnormal bleeding. Approximately 80-90% of bleeding episodes occur in the musculoskeletal system, especially in the large synovial joints and muscles. Repeated haemarthrosis induce joint cartilage damage and irreversible degenerative joint disease.

Regular intravenous administration of coagulation factor concentrates starting after the first joint bleed and/or before the age of 2 ('primary' prophylaxis) is now the evidence-based, first-choice treatment in children with severe haemophilia. This primary prophylaxis has radically decreased the incidence of arthropathy in patients with haemophilia. Despite the positive effect of primary prophylaxis on arthropathy at several joints, the ankle joint seems to be an exception to the rule, as patients with haemophilia treated with primary prophylaxis still experience ankle arthropathy. As such, the ankle now is the main affected joint in patients with haemophilia under the age of 20. This makes the scientific community facing a new challenge. Determining aetiologic/contributing factors associated to the ankle arthropathy pathophysiological cascade in children with haemophilia (CwH) is therefore a primary objective in the haemophilic research community nowadays.

Loading of the ankle is crucial as the ankle plantar flexors provide the main propulsive power during gait, the tibiotalar joint caries a complex distribution of joint stresses as a consequence of talar morphology and kinematics and, from a biomechanical and biochemical viewpoint, differs significantly from other major lower limb joints. Previous biomechanical studies focused on kinematic and strength measures, however, they omitted to incorporate fundamental measures of joint loading (joint kinetics) and joint structural integrity (JSI, assessment of soft tissue and osteochondral integrity through MRI). This makes it impossible to draw firm conclusions on biomechanical contributing factors. Furthermore, few, low-quality studies focused on conservative treatment strategies (e.g. strength training, mobilisation, proprioceptive training) in patients with ankle arthropathy. In a minority of the cases, important adverse effects (joint bleeding during strength and proprioception training) have been reported. Because of the low quality of the intervention studies and the lack of biomechanical studies focusing on joint loading and joint integrity, it is impossible to pinpoint the aetiology of these side effects. One assumption might be that side effects originate from inappropriate conservative approaches as a consequence of lacking knowledge on joint loading and joint integrity.

An innovative approach within the domain of ankle arthropathy in CwH is therefore to study foot and lower limb kinetics during gait. The quantification of foot joints kinetics encompasses considerable challenges and, until recently, only simplified single-segment foot models have been used. Those models typically underestimate the mechanical contribution of the different foot joints and, of equal importance, overestimate the kinetic contribution of the tibiotalar joint.

To overcome the above mentioned shortcomings, a valid 3D Multisegment Foot Kinetic Model (3DMFKM) should be developed and introduced within the population of CwH. This is important as it allows to quantify increased loading at the tibiotalar joint (or other joints) that may help to explain this ankle arthropathy in these patients. This will have been missed by previous research due to the consideration of the foot as one entire segment.

Providing a classification system based on these kinetic data would, in a second stage, be a pertinent and valuable approach as this provides a rationale for designing randomized controlled trials.

In this perspective, it is also recommended to assess the relationship with other biomechanical and anatomical determinants, especially if one aims at developing optimal management and rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Aged range 6-18 years
* All levels of severity of haemophilia A or B, and on all types of treatment.

Exclusion Criteria:

* Excluded will be those with an acute bleed within 12 weeks prior to testing and those with an uncontrolled high titre inhibitor.

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with haemophilia
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Kinetic Joint Classification System outcome measure | month 24
  Kinetic Joint classification system encompasses a classification system based on mechanical loading profiles of foot joints measured during barefoot walking

SECONDARY OUTCOMES:
Instrumentation implementation outcome measure | month 12
  Before the Kinetic Joint Classification System can be developed, a number of technical challenges needs to be tackled. Thus, this outcome measure reflects the adequate implementation of measurement technology for assessing gait pattern and mechanical loading of foot joints during walking
MRI and Haemophilia Joint Health Score correlation outcome measure | month 24